CLINICAL TRIAL: NCT06509854
Title: PAthwAy of Dyspneic patIent in Emergency in France
Acronym: Fr-PArADIse
Status: Not yet recruiting | Type: Observational
Sponsor: Pr. Nicolas GIRERD (Other)
Responsible Party: Sponsor-Investigator, Pr. Nicolas GIRERD, Clinical Professor, Central Hospital, Nancy, France
Organization: Central Hospital, Nancy, France (Other)
Other Study IDs: 2022PI21
Record Dates: First submitted 2024-07-04; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Acute Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational retrospective multi-center study focuses on patients treated for acute dyspnea by emergency medical teams. The primary objective is to identify factors associated with the risk of mortality and rehospitalization in these patients. This evaluation will be conducted both overall and within specific subgroups of interest, including gender (men/women), age categories, mode of admission, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Man or women aged 18 years and older.
* Patients with acute dyspnea managed by a medical emergency team at the investigator centers between 2010 and 2021.

Exclusion Criteria:

- Cardiorespiratory arrest before emergency department management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated in the emergency department for acute dyspnea.
Sampling Method: Non-Probability Sample
Enrollment: 89700 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
All-cause post-hospitalization mortality and rehospitalization | Within 5 years following hospital discharge
  Composite endpoint of all-cause post-hospitalization mortality and rehospitalization

SECONDARY OUTCOMES:
Proportion of readmissions (all-cause and specific - including hospitalization for acute dyspnea ). | 1 month and 1 year post admission for acute dyspnea in the emergency department
Post admission mortality | Within 20 years following hospital discharge
  Assessed by: Composite criterion of rehospitalization and/or death following emergency department admission (short and long-term). with outcome 5.
Post admission rehospitalization | Within 20 years following hospital discharge
  Assessed by: Composite criterion of rehospitalization and/or death following emergency department admission (short and long-term) with outcome with outcome 4.
Erroneous etiological diagnosis of dyspnea in the emergency department | Within hospital stay, maximum 21 days
  Assessed by: defined as a discrepancy between the diagnosis at discharge from the emergency department and the final diagnosis in the hospital discharge letter
All-cause mortality and specific mortality (cardiovascular and non-cardiovascular). | Within 5 years following hospital discharge
  Assessed by: Composite endpoint of all-cause mortality and specific mortality (cardiovascular and non-cardiovascular) with outcome 8
Emergency post-admission mortality | Within 20 years following hospital discharge
  Assessed by: Composite criterion of mortality and rehospitalization post-admission for acute dyspnea in the emergency department over the long term with outcome 9
Emergency post-admission rehospitalisation | Within 20 years following hospital discharge
  Assessed by: Composite criterion of mortality and rehospitalization post-admission for acute dyspnea in the emergency department over the long term outcome 8
Duration of stay in the emergency department | Within hospital stay, maximum 21 days
  Assessed by: Duration of stay in the emergency department
Erroneous etiological diagnosis of dyspnea in the emergency department | Within hospital stay, maximum 21 days
  Assessed by: Erroneous etiological diagnosis of dyspnea in the emergency department
In-hospital mortality | Within hospital stay, maximum 21 days
  Assessed by: In-hospital mortality
Length of hospital stay | Within hospital stay, maximum 21 days
  Assessed by: Length of hospital stay
Post emergency admission (For dyspnea) mortality and rehospitalization | Within 5 years following hospital discharge
  Assessed by: Post emergency admission (For dyspnea) mortality and rehospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Tahar CHOUIHED, MD, PhD, Principal Investigator — Central Hospital, Nancy, France; Nicolas GIRERD, MD, PhD, Principal Investigator — CHRU de Nancy
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - CHU de Dijon, Dijon
  - Hospices civils de Lyon, Groupement Hospitalier Édouard-Herriot, Lyon
  - CHRU of Nancy, Nancy